CLINICAL TRIAL: NCT00286910
Title: Urinary Aquaporin 2 and Expression of the NPHS2 Gene in Adults Suffering From Nephrotic Syndrome
Status: Completed | Type: Observational
Sponsor: Regional Hospital Holstebro (Other)
Responsible Party: Holstebro Hospital, Erling Bjerregaard Pedersen
Other Study IDs: MED.RES.HOS.2005.05/ IMT
Record Dates: First submitted 2006-02-03; First posted 2006-02-06 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2010-03

CONDITIONS: Nephrotic Syndrome
Keywords: AQP-2; NPHS2-gene
MeSH Terms: conditions — Nephrotic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

SUMMARY:
We want to test the hypothesises that patients with nephrotic syndrome have a higher excretion of AQP2 in the urine,that they have a higher concentration of AVP,and a lower C-H2O.Everything will normalize, when the syndrome is in remission.Furthermore we want to test the hypothesis that the expression of mutations in the NPHS2-gene,that codes for podocin,will cause a lack off or a poorer response in the treatment of nephrotic syndrome

ELIGIBILITY:
Inclusion Criteria:

adult patients with nephrotic syndrome in the years 1995 until now; both male and female; the kidney disease must be based upon a kidney biopsy ; age > 18 years -

Exclusion Criteria:

severe diseases in the heart, lungs or liver; diabetes mellitus; other not well-treated diseases in endocrine organs; cancer unwillingness to participate

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adult patients with nephrotic syndrome healthy volunteers
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2005-05

CONTACTS AND LOCATIONS:
Overall Officials: Erling B Pedersen, professor, Study Chair — Holstebro Hospital, Denmark
Locations (1):
- Department of Medicine, Holstebro Hospital, Holstebro, Denmark